CLINICAL TRIAL: NCT05772624
Title: Safety and Efficacy Evaluation of Low-dose Nivolumab in Combination With AVD as Frontline Therapy for Classic Hodgkin's Lymphoma
Brief Title: Lowdose Nivolumab in Combination With AVD as Front Line Therapy for Classic Hodgkin's Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitario Dr. Jose E. Gonzalez (Other)
Responsible Party: Principal Investigator, David Gomez Almaguer, Dr., Hospital Universitario Dr. Jose E. Gonzalez
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HE23-0001
Record Dates: First submitted 2023-02-13; First posted 2023-03-16 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Safety Issues; Efficacy, Self
Keywords: Nivolumab; lowdose nivolumab; NAVD; hodgkin's lymphoma
MeSH Terms: conditions — Hodgkin Disease | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- LowN-AVD (Experimental): classic Hodgkin's lymphoma patients receiving low dose nivolumab in combination with AVD
  Interventions: Drug: low dose nivolumab in combination with AVD

INTERVENTIONS:
Drug: low dose nivolumab in combination with AVD — Nivolumab as an standard dose of 40mg in combination with AVD.

SUMMARY:
This study aims to prove the efficacy and safety of low dose nivolumab (40mg as the lowest available presentation) in combination with AVD (adriamycin,vinblastine sulfate and dacarbazine) as frontline treatment for classic Hodgkin's lymphoma.

DETAILED DESCRIPTION:
The main objective of this project is to prove the efficacy and safety of Nivolumab used as an standard dose of 40mg ( as the lowest available presentation) in combination with AVD as frontline therapy for Hodgkin's lymphoma.

Patients classification.

We will categorize patients in three groups as follows:

1. Early stages by Ann-arbor classification (I,II) with no risk factors (as stablished by NCCN's guidelines criteria).
2. Early stages by Ann.arbor classification (I,II) with risk factors ( as stablished by NCCN's guidelines criteria).
3. Advanced stages by Ann-arbor classification (III,IV).

Methodology:

* Patients will receive two initial cycles of NAVD therapy ( each with two applications in day 1 and 15) and then will be evaluated with an interim PET/CT after completing cycle 2.
* According to the PET C/T results, patients will be categorized as fast responsers (patients who achieve Deauville 1-3 classification) and low responsers ( patients who achieve Deauville 4-5).
* Fast responsers will receive following cycles without nivolumab (2 extra cycles for patients categorized as early stage with no risk factors, 4 extra cycles for patients categorized as early stages with risk factors and for advanced stages).
* Patients will receive medical evaluation at first meeting, during their treatment and after conclusion of the treatment with physical examination and laboratory tests according to medical criteria.
* Adverse effects will be recorded and managed following the guidelines for immunotherapy and chemotherapy indications.

ELIGIBILITY:
Inclusion Criteria:

* Patients with recent diagnosis of classic Hodgkin's lymphoma demonstrated by incisional or excisional biopsy of adenopathy.
* Treatment naive patients.
* Any stage
* Any functional status.

Exclusion Criteria:

* Patients with refractory or relapsed disease.
* Patients with non classical variety.
* Patients with chronic or active infections at the moment of recruiting.
* Patients younger than 16 years old.
* Pregnancy

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2023-02-13 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
To determine general response | Six weeks after completion of therapy.
  To determine patients achieving either a complete response or a partial response as demonstrated with PET C/T evaluation.

SECONDARY OUTCOMES:
Response duration | up to 2 years
  To evaluate the duration of the response achieved with the therapy.
Adverse effects | through the study completion and up to 6 months
  To record the side effects associated with the treatment as stablished by the international guidelines for chemotherapy and immunotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Perla R Colunga Pedraza, MD, Principal Investigator — Hospital Universitario Jose Eleuterio Gonzalez
Locations (1):
- Hospital Universitario Dr Jose Eleuterio Gonzalez, Monterrey, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hwang YY, Khong PL, Kwong YL. Low-dose nivolumab induced remission in refractory classical Hodgkin lymphoma. Ann Hematol. 2017 Jul;96(7):1219-1220. doi: 10.1007/s00277-017-3007-9. Epub 2017 Apr 22. No abstract available. PMID 28434018
- [Result] Lepik KV, Fedorova LV, Kondakova EV, Zalyalov YR, Babenko EV, Lepik EE, Kotselyabina PV, Beynarovich AV, Popova MO, Volkov NP, Stelmakh LV, Baykov VV, Moiseev IS, Mikhailova NB, Kulagin AD, Afanasyev BV. A Phase 2 Study of Nivolumab Using a Fixed Dose of 40 mg (Nivo40) in Patients With Relapsed/Refractory Hodgkin Lymphoma. Hemasphere. 2020 Sep 23;4(5):e480. doi: 10.1097/HS9.0000000000000480. eCollection 2020 Oct. PMID 33062947
- [Result] Brockelmann PJ, Goergen H, Keller U, Meissner J, Ordemann R, Halbsguth TV, Sasse S, Sokler M, Kerkhoff A, Mathas S, Huttmann A, Bormann M, Zimmermann A, Mettler J, Fuchs M, von Tresckow B, Baues C, Rosenwald A, Klapper W, Kobe C, Borchmann P, Engert A. Efficacy of Nivolumab and AVD in Early-Stage Unfavorable Classic Hodgkin Lymphoma: The Randomized Phase 2 German Hodgkin Study Group NIVAHL Trial. JAMA Oncol. 2020 Jun 1;6(6):872-880. doi: 10.1001/jamaoncol.2020.0750. PMID 32352505
- [Result] Chan TSY, Hwang YY, Khong PL, Leung AYH, Chim CS, Tse EWC, Kwong YL. Low-dose pembrolizumab and nivolumab were efficacious and safe in relapsed and refractory classical Hodgkin lymphoma: Experience in a resource-constrained setting. Hematol Oncol. 2020 Dec;38(5):726-736. doi: 10.1002/hon.2787. Epub 2020 Aug 20. PMID 32786092
- [Result] Ramchandren R, Domingo-Domenech E, Rueda A, Trneny M, Feldman TA, Lee HJ, Provencio M, Sillaber C, Cohen JB, Savage KJ, Willenbacher W, Ligon AH, Ouyang J, Redd R, Rodig SJ, Shipp MA, Sacchi M, Sumbul A, Armand P, Ansell SM. Nivolumab for Newly Diagnosed Advanced-Stage Classic Hodgkin Lymphoma: Safety and Efficacy in the Phase II CheckMate 205 Study. J Clin Oncol. 2019 Aug 10;37(23):1997-2007. doi: 10.1200/JCO.19.00315. Epub 2019 May 21. PMID 31112476